CLINICAL TRIAL: NCT05902845
Title: Efficacy, Safety and Cytopharmacokinetics of RD13-02 Cell Injection in the Treatment of Patients With Recurrent or Refractory CD7-positive Hematologic Malignancies
Brief Title: RD13-02 CAR-T Cell Injection for Patients With r/r CD7+ T-ALL/T-LBL
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Xiaoyu Zhu (Other Government)
Collaborators: Nanjing Bioheng Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Xiaoyu Zhu, Clinical Professor, Anhui Provincial Hospital
Organization: Anhui Provincial Hospital (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BHCT-RD13-02-08
Record Dates: First submitted 2023-05-23; First posted 2023-06-15 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Neoplasms; Hematologic Neoplasms; Hematologic Diseases
MeSH Terms: conditions — Neoplasms; Hematologic Neoplasms; Hematologic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RD13-02 cell infusion (Experimental): drugs use generic name : RD13-02 CAR-T cell injection; dosage form : Cell injection dosage : 2×10^8 CAR+ T cells frequency : Once
  Interventions: Drug: RD13-02 cell infusion

INTERVENTIONS:
Drug: RD13-02 cell infusion — CAR-T cells

SUMMARY:
This is a single-arm, open-label, single-center, phase I study. The primary objective is to evaluate the safety of CD7 CAR-T therapy for patients with CD7-positive relapsed or refractory T-ALL/LBL, and to evaluate the pharmacokinetics of CD7 CAR-T in patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age 3-70
2. Diagnosis of r/r T-ALL/LBL.
3. CD7 positive expression
4. Bone marrow lymphoblasts ≥5% by morphologic evaluation at screening
5. Creatinine clearance (as estimated by Cockcroft Gault) ≥ 60 mL/min, Serum alanine aminotransferase(ALT)/aspartate aminotransferase(AST) < 3×upper limit of normal, Total bilirubin < 1.5×upper limit of normal or ≤1.5mg/dl
6. Left ventricular ejection fraction ≥ 50% .
7. Baseline oxygen saturation ≥ 92% on room air.
8. ECOG performance status of 0 to 2.
9. The estimated survival time is more than 3 months.
10. Subjects or their legal guardians volunteer to participate in the study and sign the informed consent.

Exclusion Criteria:

1. Sujects with concomitant genetic syndromes associated with bone marrow failure states.
2. Sujects with some cardiac conditions will be excluded.
3. History of traumatic brain injury, consciousness disturbance, epilepsy, cerebrovascular ischemia, and cerebrovascular hemorrhagic disease, which might compromise the ability of the subject to compliance with the obligations under the protocol.
4. History of malignancy other than non-melanoma skin cancer or carcinoma.
5. Primary immune deficiency.
6. Presence of uncontrolled infections.
7. Sujects with some anticancer therapy before CAR-T infusion will be excluded.
8. Active uncontrolled acute infections.
9. Known history of infection with human immunodeficiency virus (HIV); active or latent hepatitis B, hepatitis C and syphilis.
10. Subjects who are receiving systemic steroid therapy prior to screening.
11. Subjects with acute graft-versus-host disease (GvHD)
12. Having received live/attenuated vaccine within 4 weeks prior to screening.
13. History of allergy to any component of the cell therapy product.
14. Pregnant or breastfeeding women
15. Any other issue which, in the opinion of the investigator, would make the sujects ineligible for the study.

Ages: 3 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2023-04-30 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Overall response rate, ORR | Evaluate at 4 weeks after CAR-T infusion
  The proportion of patients with CR (complete response) /CRi (complete response with incomplete blood cell recovery) and PR (partial response).
Overall response rate, ORR | Evaluate at 8 weeks after CAR-T infusion
  The proportion of patients with CR (complete response) /CRi (complete response with incomplete blood cell recovery) and PR (partial response).
Overall response rate, ORR | Evaluate at 12 weeks after CAR-T infusion
  The proportion of patients with CR (complete response) /CRi (complete response with incomplete blood cell recovery) and PR (partial response).

SECONDARY OUTCOMES:
Overall response rate with MRD-negative, MRD-ORR | Up to 1 years after CAR-T infusion
  Proportion of patients achieving CR/CRi who is MRD-negative in bone marrow
Duration of remission, DOR | Up to 1 years after CAR-T infusion
  The time from CR/CRi and PR to disease relapsed or death due to disease progression after CAR-T infusion
Event-free survival, EFS | Up to 1 years after CAR-T infusion
  The time from first achieving CR/CRi to relapse or death
The proportion of patients who receive hematopoietic stem cell transplantation | Up to 1 years after CAR-T infusion
  The proportion of subjects who achieved remission after infusion who received HSCT.
Overall survival, OS | Up to 1 years after CAR-T infusion
  The time from CAR-T infusion to death due to any cause

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of University of Science and Technology of China, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No